CLINICAL TRIAL: NCT00412243
Title: Phase I/II Study of Clofarabine Plus Cyclophosphamide for Relapsed and Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Clofarabine and Cyclophosphamide Combination in Acute Lymphoblastic Leukemia Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0552
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Burkitt's Lymphoma; Lymphoblastic Lymphoma; Acute Lymphoblastic Leukemia
Keywords: Burkitt's Lymphoma; Lymphoblastic Lymphoma; Acute Lymphoblastic Leukemia; Clofarabine; Clofarex; Clolar; Cyclophosphamide; Neosar; Cytoxan
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine + Cyclophosphamide (Experimental): Clofarabine 40 mg/m^2 daily for 3 Days + Cyclophosphamide starting 200 mg/m^2 every 12 hours for 3 days
  Interventions: Drug: Clofarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Clofarabine — 40 mg/m^2 Daily for 3 Days
  Other Names: Clorarex; Clolar
Drug: Cyclophosphamide — Beginning dose 200 mg/m^2 every 12 hours for 3 days
  Other Names: Cytoxan; Neosar

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the drugs clofarabine and cyclophosphamide that can be given together in the treatment of relapsed or refractory ALL. The safety of the combination treatment will also be studied.

Objectives:

Phase I:

1. To establish toxicities and safety of the proposed combination
2. To establish the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of the combination to proceed with the phase II part of the study

   Phase II:
3. To establish the efficacy (complete and overall response) of the proposed combination.
4. To analyze pharmacokinetic (PK) and pharmacodynamic (PD) properties of clofarabine as well as the impact on DNA repair of leukemic blasts with the proposed combination.

DETAILED DESCRIPTION:
Clofarabine is a drug that is designed to interfere and disrupt important metabolic pathways of cancer cells by interfering with their multiplication and slowing or stopping their growth. Cyclophosphamide is also designed to destroy cancer cells by interfering with their multiplication and slowing or stopping their growth and spread throughout the body. Cyclophosphamide is commonly used in the treatment of ALL.

If you are found to be eligible to take part in this study, you will receive clofarabine by vein over about 60 minutes, once a day for 3 to 5 days. Cyclophosphamide will be given by vein over about 3 hours, twice a day for 3 to 5 days. These 3-5 days are considered 1 cycle of therapy.

As the safety of this combination has not been established yet, at least the first 2 participants on this study will receive clofarabine for 3 days and cyclophosphamide at a lower dose than usually given for 3 days (6 doses). Should there be no serious side effects that can be related to the study drugs, the next group of 2 participants will receive clofarabine over 3 days and a slightly higher dose of cyclophosphamide for 3 days (6 doses). Should there still be no serious side effects at that level, 2 further levels will be tested where both clofarabine and cyclophosphamide are then given over 4 days and eventually 5 days. Should serious and study drug-related side effects occur at any point during this increase of doses, a certain dose level along this increase will be defined as the appropriate dose for all future participants to receive. It is estimated that about 30 participants will receive therapy during the dose escalations portion of this study (Phase I). It is estimated that about 25 more participants will receive therapy at the dose levels that are considered best (Phase II).

During treatment, you will have a physical exam at least once a week. You may also be asked about the level of your daily activities, how you are feeling, and which medications you are taking currently. Routine blood samples (about 1 tablespoon each) will be drawn at least 1-3 times weekly and more frequently if considered necessary. A bone marrow aspirate and/or biopsy will be repeated starting at about Day 14 and will be repeated every 1 to 2 weeks until the study doctors can decide for sure whether you have responded or not. In some cases, a repeat bone marrow test may not be necessary, but this decision will be made by your treating doctor.

If you respond well after your first round of therapy, you may receive up to 6 additional courses of therapy. Each course will be repeated about every 3 to 7 weeks at a slightly lower dose of both drugs than was used during the first round of therapy. Later doses can also be changed depending on what type of side effects you may experienced with earlier rounds of therapy.

At the end of the study, a heart scan (either an Echo or MUGA scan) will be repeated. About 1 tablespoon of blood will be taken for routine blood tests. A focused physical exam may also be repeated.

This is an investigational study. All drugs in this study are FDA approved and commercially available. Their use together in this study is investigational. . About 55 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated ALL (including Burkitt's lymphoma and lymphoblastic lymphoma) in relapse or primary refractory. For patients in first relapse, the first remission duration may not exceed 12 months.
2. Age >/= 21 years.
3. Zubrod performance status </= 3.
4. Adequate liver function (bilirubin </= 2.5 mg/dL and Serum glutamic pyruvic transaminase (SGPT or SGOT) </= 3 * ULN, unless considered due to tumor), and renal function (glomerular filtration rate [GFR] >/= 60 mL/min). Even if organ function abnormalities are considered due to tumor, the upper limit for bilirubin is </= 5 mg/dL and creatinine </= 3 mg/dL.
5. Male and female patients who are fertile agree to use an effective barrier method of birth control (e.g., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 14 days of study enrollment (applies only if patient is of childbearing potential. Non-childbearing is defined as >/= 1 year postmenopausal or surgically sterilized).

Exclusion Criteria:

1. Patients with active heart disease (New York Heart Association (NYHA) class >/= 3 as assessed by history and physical examination).
2. Patients with a cardiac ejection fraction (as measured by either Multi Gated Acquisition Scan (MUGA) or echocardiogram) < 45% are excluded.
3. Patients who receive other chemotherapy. Patients must have been off previous therapy for >/= 2 weeks and must have recovered from acute toxicity of all previous therapy prior to enrollment. (Concurrent therapy for central nervous system (CNS) prophylaxis or treatment for CNS relapse is permitted). Treatment may start earlier if necessitated by the patient's medical condition following discussion with the Principal Investigator.
4. Pregnant and breast-feeding patients are excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 3/21/2006 - 3/3/2011; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: One enrolled participant was excluded.
Groups:
- Clofarabine + Cyclophosphamide: Clofarabine 40 mg/m^2 daily for 3 Days + Cyclophosphamide starting 200 mg/m^2 every 12 hours for 3 days
  Clofarabine : 40 mg/m^2 Daily for 3 Days
  Cyclophosphamide : Beginning dose 200 mg/m^2 every 12 hours for 3 days
Period: Overall Study
Arm/Group | Clofarabine + Cyclophosphamide
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 50
Age Continuous [Median (Full Range); unit: years] | 30 [21 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose for Cyclophosphamide (MTD)
Description: MTD is dose at which there are no dose limiting toxicity (DLT) defined as any =/> grade 3 drug-related non-hematologic toxicity that occurs within the first 14 days after start of treatment. Evaluation using continual reassessment method; 3-5 Day Cycle
Time Frame: First 14 days of each cycle
Population: MTD calculated with first 8 study participants.
Measure: Number; unit: mg/m^2
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 8
mg/m^2 | 200

ADVERSE EVENTS:
Time Frame: Six years
Arm/Group | Clofarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cyclophosphamide (N=50)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 8 (8)
Elevated Amylase (Blood and lymphatic system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Infection (Infections and infestations) | 4 (4)
Elevated Lipase (Blood and lymphatic system disorders) | 1 (1)
Hyperbiliruninemia (Hepatobiliary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cyclophosphamide (N=50)
Nausea/Vomiting (Gastrointestinal disorders) | 39 (44)
Dairrhea (Gastrointestinal disorders) | 16 (18)
Stomatitis/Mucositis (Gastrointestinal disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 17 (17)
Elevated Liver Function Tests (Hepatobiliary disorders) | 25 (25)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No